CLINICAL TRIAL: NCT05371301
Title: Efficacy of Primary Debulking Surgery Versus Neoadjuvant Chemotherapy in Stage IV Ovarian Cancer: a Phase III Randomized Controlled Study
Brief Title: Efficacy of Primary Debulking Surgery Versus Neoadjuvant Chemotherapy in Stage IV Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-GYN-20200816
Record Dates: First submitted 2022-04-28; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Neoadjuvant Chemotherapy; Interval Debulking Surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — CP protocol; Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NACT-IDS (Experimental): For patients whoes WB-DWI/MRI Suidan Standard Evaluation≥4 Neoadjuvant chemotherapy: platinum-based combination regimen 3 courses
  Interventions: Drug: Paclitaxel, Carboplatin; Procedure: debulking surgery
- PDS (Active Comparator): For patients whoes WB-DWI/MRI Suidan Standard Evaluation<4
  Interventions: Procedure: debulking surgery

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin — Paclitaxel 175mg/m2 iv d1 followed by Carboplatin(AUC=5) iv d1
  Arms: NACT-IDS
Procedure: debulking surgery — Remove all visible tumors and any other tissues or organs where tumor may have spread, which may include:
  Uterus Fallopian tubes Omentum (tissue that covers the stomach, large intestine and other abdominal organs) Lymph nodes Diaphragm Part of the large bowel Spleen Parts of the liver

SUMMARY:
Epithelial ovarian cancer is mostly diagnosed at late stage (III/IV), and the standard treatment for ovarian cancer includes primary debulking surgery and platinum-based adjuvant chemotherapy. However, scholars suggest that neoadjuvant chemotherapy can be used to reduce the tumor load and control the patient's condition. The aim of this study is to verify the efficacy of primary debulking surgery versus neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) is one of the most common malignant tumors in women. Due to the insidious onset and the lack of effective early diagnosis measures, about 70% of patients with epithelial ovarian cancer are already in FIGO stage III-IV at the time of diagnosis. With extensive tumor dissemination and metastasis, the 5-year survival rate of EOC patients is only about 30-40%.

Currently, the standard treatment for ovarian cancer remains to include primary debulking surgery(PDS) and platinum-based adjuvant chemotherapy. Despite the lack of evidence from prospective randomized controlled studies, evidence invariably shows that satisfactory debulking surgery improves survival prognosis in advanced ovarian cancer and that this benefit is significantly associated with the amount of residual lesion.

How to increase the proportion of patients with satisfactory tumor reduction (residual lesions <1 cm) has long been a pressing issue for gynecologic oncologists. However, because ovarian cancer lesions are mainly disseminated in the pelvic cavity, the extent of surgery to achieve satisfactory reduction is often large and difficult to be tolerated for some patients. At the same time, due to the large initial tumor or the limited treatment level, some patients are unable to obtain satisfactory cytoreduction. Therefore, some scholars suggest that neoadjuvant chemotherapy (NACT) can be used to reduce the tumor load and control the patient's condition, followed by interval debulking surgery (IDS), called NACT-IDS treatment model.

Whether the NACT-IDS treatment model can be used as a conventional alternative to PDS has been controversial. The foundation for NACT-IDS was laid by two multicenter randomized controlled phase III clinical trials, EORTC 55971 and CHORUS. Both studies showed that the application of NACT in patients with advanced ovarian cancer resulted in a higher proportion of satisfactory cytoreduction and lower postoperative complications and mortality while ensuring a similar prognosis. However, the two studies mentioned above have been questioned by some scholars because of the lower median operative time, lower percentage of satisfactory cytoreduction, and lower patient prognosis than the international general level. Meanwhile, another phase III randomized controlled clinical trial, JCOG0602, was a non-inferiority trial, and the results did not confirm that NACT was not inferior to PDS. Therefore, at present, NCCN guidelines recommend that PDS remains the first choice for most patients.

At present, there are no relevant clinical trials comparing the impact of PDS with NACT on the prognosis of patients with ovarian cancer. In this study, investigators propose to assess the resectability of patients with abdominopelvic lesions using the Suidan standard resectability prediction model based on the evaluation of WB-DWI/MRI. In patients of stage IV ovarian cancer with resectable abdominopelvic lesions, the prognostic impact of PDS and NACT will be compared prospectively and randomly, with the aim of providing a new decision basis for the treatment of patients with stage IV ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years of age.
* ECOG 0-2
* Clinically confirmed epithelial ovarian or fallopian-tube cancer or primary peritoneal cancer
* FIGO2014 stage III/IV
* Sign the informed consent form
* Good compliance and agree to cooperate with survival follow-up

Exclusion Criteria:

* Patients with large abdominal masses or other reasons for not being able to tolerate surgical treatment
* Patients with severe medical comorbidities that cannot be corrected in the short term and are not suitable for tumor cytoreductive surgery
* Patients with contraindications to chemotherapy
* Patients with a history of psychotropic substance abuse and unable to quit or patients with mental disorders
* Patients with serious safety hazards or concomitant diseases that, in the judgment of the institution, would affect the patient's ability to complete the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | 5 year
  Patients from surgery or neoadjuvant chemotherapy to disease progression or time to last follow-up
overall survival | 5 year
  Patients from surgery or neoadjuvant chemotherapy to death or time to last follow-up

OTHER OUTCOMES:
postoperative residual lesions | during surgery
  R0: no residue under the microscope after resection R1: residue≤1cm R2: tumor residue visible to the naked eye(>1cm)
platinum sensitivity | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, PhD&MD, Principal Investigator — Fudan university shanghai cancer center, Deparment of gynecologic oncology
Locations (1):
- Fudan university shanghai cancer center, Deparment of gynecologic oncology, Shanghai, Shanghai Municipality, China